CLINICAL TRIAL: NCT06169111
Title: REGulatory T Cells in Autism Induced by Maternal Immune Activation
Acronym: REGAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230622; IDRCB: 2023-A01329-36 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2023-11-24; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: neurodevelopemental disorders; immunology; regulatory T lymphocytes
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Spectrum Disorders (ASD) patients with Maternal Immune Activation (MIA) (Experimental)
  Interventions: Biological: REGulatory T cells in Autism induced by maternal Immune activation
- Autism Spectrum Disorders (ASD) patients without Maternal Immune Activation (MIA) (Active Comparator)
  Interventions: Biological: REGulatory T cells in Autism induced by maternal Immune activation

INTERVENTIONS:
Biological: REGulatory T cells in Autism induced by maternal Immune activation — REGulatory T cells in Autism induced by maternal Immune activation

SUMMARY:
Autism Spectrum Disorders (ASD) represent a heterogeneous clinical entity of neurodevelopmental disorders affecting around 1% of the general population (Lord et al. 2020). There is currently no curative treatment for patients with ASD, and management does not take into account the existence of specific patient subgroups. Beyond genetic factors (Delorme et al. 2013), environmental factors play a fundamental role in the determinism of ASD. Among them, maternal immune activation (MIA) during pregnancy is a recognized risk factor for ASD in children (Estes and McAllister 2016). Our team has helped to demonstrate that MIA induced by infections or autoimmune pathologies in the mother during pregnancy (particularly at the end of the 1st trimester/beginning of the 2nd trimester) significantly increases the risk of ASD in the offspring (Antoun et al. 2021). Mechanistically, MIA leads to a deregulation of the regulatory T lymphocyte (Tregs)/Th17 balance (in the direction of a decrease in anti-inflammatory Tregs and an increase in pro-inflammatory Th17) in the mother but also, via epigenetic mechanisms, in the fetus (Lim et al. 2021). Our team have recently demonstrated the same Tregs/Th17 deregulation profile in ASD patients (Ellul et al. 2021). This disruption of the Tregs/Th17 balance is responsible for disrupting fetal brain development via IL-17 receptors present on fetal neurons (Choi et al. 2016). Importantly, these socio-communicative and morphological abnormalities appear, in specific animal models, to be reversible upon restoration of the Tregs/Th17 balance (Z. Xu et al. 2021; Choi et al. 2016). While data on the involvement of IL-17 are becoming better known, the role of Tregs in this model has been surprisingly little studied.Our overall aim is therefore, in humans and mice, to determine the role of Tregs and IL-17-producing lymphocytes in the development and maintenance of autistic symptoms triggered by MIA.

Our specific objectives in humans will be to use an existing cohort (EXPECT) of ASD patients to compare those with and without a history of MIA using a standardized clinical evaluation (including overall autism severity, language and motor development, adaptive behaviors,comorbidities), a systems immunology assessment (combining deep immunophenotyping by flow cytometry, cytokine measurements - simultaneous Luminex assay of 50 pro-inflammatory cytokines associated with Th1/Th2/Th17/Treg responses) and a targeted quantitative metabolomics analysis of the tryptophan pathway.

DETAILED DESCRIPTION:
The aim of the REGAIN project will be to study in detail the cellular populations involved in the development of MIA-mediated autistic symptoms in humans.

Based on both our preliminary meta-analysis data and previous work on Tregs work on Tregs, our team calculated that the number of subjects needed to meet our primary objective on Tregs was (with risk α = 0.05, power power 1 - β =0.9 and a minimum detectable odds ratio = 5) of 30 patients per group (3.75 p/month for 24 months).

The Center of Excellence for Autism and Neurodevelopmental Disorders (InovAND) at Robert Debré Hospital receives around 500 new ASD patients a year (40p/month). Furthermore, in humans, it is estimated that 15% of autisms could be linked to an ASI. Over the period of our study, this should represent around 75 patients/year (7p/month) at Robert Debré. For safety reasons, to include enough patients but taking into account the drop in activity due to the COVID-19 crisis, our team decided to include decided to include 35 patients/group (4.37 p/month for 24 months = 1.45 p/month/group).

During hospitalization for the diagnostic workup at InovAND (Robert Debré hospital), and as part of the care provided, patients will be assessed by psychiatrists specializing in autism who will take a family history, ascertain the presence or absence of MIA, collect the child's personal and neurodevelopmental history, and obtain parental consent for inclusion in the cohort. Psychologists, speech therapists and psychomotor therapists will then assess the patients using the standardized scales described above. If the parents have given their consent to participate in REGAIN, the patients will have a sample taken for the purposes of the research. blood sample at the end of the clinical evaluation.

As part of standard care, each child will benefit from a standardized assessment based on (i) autism reference interviews; the Social Reciprocity Scale (SRS); (ii) the Autism Diagnostic Interview (ADI) Autism Diagnostic Observation (iii) assessment of general cognitive abilities and adaptive behavior profile (Wechsler scales or Raven's progressive matrices for non-verbal individuals, Vineland II scale); (iv) a special effort will be made to characterize the main symptoms of autism. More specifically, repetitive behaviors and sensory abnormalities will be explored using the Repetitive Behavior Scales (revised version) and Dunn's Sensory Profile. (v) Psychiatric and somatic comorbidities associated with immune dysregulation will also be explored (ADHD, chronic tics frequently reported in PANS syndrome, gastrointestinal symptoms, immunoallergic comorbidities) using a semi-structured interview our team have constructed.

Characterization of maternal history of MIA: Due to the intrinsic nature of our study design, Our team will not be able to prospectively explore ASI during pregnancy in mothers. Therefore, our team will include patients in the MIA+ category if their mother had a significant history suggestive of MIA during pregnancy.

As previously mentioned, the children included in REGAIN are part of a larger cohort of children with ASD (also including healthy controls) followed at the Robert Debré Hospital (EXPECT and C0733 studies), for which our team already have the agreement of a French personal protection committee for the collection of clinical data and immunological samples from ASD patients (IDRCB no. IDRCB: 2021-A00489-32; Ref. CPP: 2021-27) and controls (authorization no. 917138). The purpose of this protocol and the accompanying request is to authorize the collection of fresh blood and the realization of new research objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive diagnosis of ASD according to DSM-5 (APA, 2015);
* Age at inclusion between 3 and 15 years;
* Informed consent signed by both parents and oral agreement in principle given by the subject;
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients with severe/profound intellectual disability;
* Uncontrolled epileptic seizures;
* Maternal infection during pregnancy with a pathogen with a known direct cerebral cytotoxic effect (CMV);

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare Tregs count (% CD4+) and Th17 count (% CD3+) and their ratio in ASD patients with and without MIA | 24 months
  Evaluation of the Tregs count/Th17 balance in ASD patients with and without MIA

CONTACTS AND LOCATIONS:
Overall Officials: Richard DELORME, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France